CLINICAL TRIAL: NCT03796585
Title: Assessing Barriers and Increasing Use of Immunization Registries in Pharmacies: A Randomized Controlled Trial
Brief Title: Assessing Barriers and Increasing Use of Immunization Registries in Pharmacies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tessa Hastings, Principal Investigator, Auburn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R36HS026093-01A1 (AHRQ)
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Immunization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Pharmacists assigned to this group will receive an immunization registry training program and informational flyer.
  Interventions: Behavioral: Immunization Registry Training; Behavioral: Informational flyer
- Control (Active Comparator): Pharmacists assigned to this group will receive an informational flyer. They will not receive training.
  Interventions: Behavioral: Informational flyer

INTERVENTIONS:
Behavioral: Immunization Registry Training — Education highlighting practical strategies to improve pharmacies' willingness to adopt the immunization registry and improve their ability to integrate the immunization registry into their pharmacy workflow.
  Arms: Intervention
Behavioral: Informational flyer — Informational flyer with ImmPRINT contact information

SUMMARY:
The purpose of this study is to identify barriers to utilization of immunization registries within a pharmacy context and tailor the information into a novel immunization registry training program.

DETAILED DESCRIPTION:
The purpose of this study is to identify barriers to utilization of immunization registries within a pharmacy context and tailor the information learned about barriers into a novel immunization registry training program with strategies specific to individual subsets of pharmacies, independent pharmacies in rural areas. Doing so will help achieve the long-term goal which is to increase the use of immunization registries in community pharmacies in Alabama.

The specific aims are to

1. identify barriers and best practices of immunization registry implementation,
2. use a participatory design approach to develop an immunization registry training program, and
3. disseminate and assess the impact of the immunization registry training program among community pharmacies' registry participation rates.

The impact of the training program on registry participation rates will be assessed using a randomized controlled trial design comparing Alabama community pharmacies' registry data as well as intention to participate.

ELIGIBILITY:
Inclusion Criteria:

* not currently enrolled in ImmPRINT
* currently provide at least one type of vaccination in addition to influenza
* independently owned
* agree to provide requested data for assessment

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Number of pharmacies enrolled in the Alabama Immunization Registry | 3 months
  The change in the number of participant pharmacies enrolled in the Alabama immunization registry from baseline to 3 months.

SECONDARY OUTCOMES:
Level of Immunization Registry Participation | 3 months
  Proportion of self-reported doses administered that are verified in the immunization registry.
Change in awareness | 1 month and 3 months
  The change in participant awareness of immunization registries from baseline to 3 months assessed by online questionnaire at baseline, one month, and three months. Awareness will be measured using three true or false items. Each item will be scored, 0 for an incorrect answer and 1 for a correct answer. Awareness index is the sum of the 3 items and could range from 0-3 with higher values representing greater awareness.
Change in knowledge | 1 month and 3 months
  The extent to which participant is familiar with and understands immunization registries will be assessed via online questionnaire at baseline, one month, and three months. Eight true or false and multiple answer items will be used to measure knowledge. Each item will be scored, 0 for an incorrect answer and 1 for a correct answer. Knowledge is the sum of the 8 items and could range from 0-8 with higher values representing greater knowledge.
Change in attitudes | 1 month and 3 months
  Participant's perceptions toward attributes of the immunization registry assessed via online questionnaire at baseline, one month, and three months. A scale including 25 Likert-type items will be used to measure attitudes. Each Likert-type item will be scored, ranging from 0 for strongly disagree to 6 for strongly agree. Mean scores will be calculated for the 25 items in the scale so that attitudes score range from 0 to 6 with higher values indicating greater positive attitudes.
Change in intention to enroll in immunization registry | 1 month and 3 months
  Participant's likelihood to enroll their pharmacy in the immunization registry assessed via online questionnaire at baseline and one month. A scale including 3 Likert-type items will be used to measure intention. Each Likert-type item will be scored, ranging from 0 for strongly disagree to 6 for strongly agree. Mean scores will be calculated for the three items in the scale so that intention score ranges from 0 to 6 with higher values indicating greater intention.
Change in Implementation Factors | 3 months
  Implementation factors informed by the Consolidated Framework for Implementation Research (CFIR) including innovation characteristics, characteristics of individuals, inner setting, outer setting, and process will be assessed via online questionnaire at baseline and three months. A scale including 42 Likert-type items will be used to measure Implementation Factors. Each Likert-type item will be scored, ranging from 0 for strongly disagree to 6 for strongly agree. Mean scores will be calculated so that the implementation factors score ranges from 0 to 6 with higher values indicating greater positive influence of CFIR implementation factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hastings TJ, Ha D, Fox BI, Qian J, Lakin J, Westrick SC. Increasing use of immunization information systems for routine vaccinations in independent community pharmacies: A randomized controlled trial. J Am Pharm Assoc (2003). 2022 Jul-Aug;62(4):1270-1279.e2. doi: 10.1016/j.japh.2022.02.010. Epub 2022 Feb 19. PMID 35292212